CLINICAL TRIAL: NCT04131751
Title: Establishing of Next Genaration Sequencing Methods for Microbiological Diagnostic of Ascitic Fluid Infections
Brief Title: Application of Clinical Metagenomics in the Diagnosis of Ascites
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Badr, Principal Investigator, University Hospital Freiburg
Other Study IDs: 246/19
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Ascites Infection
Keywords: Metagenomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial and fungal DNA from human ascites samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — we will investigate the sensitivity and specificity of next generation sequencing as a diagnostic tool in ascites infections.

SUMMARY:
Infection of the ascitic fluid is a serious complication associated with high morbidity and mortality. This fluid is often colonized with bacteria that can cause infection of the peritoneum and possibly sepsis. Many bacteria of the human intestinal microbiome can't be cultured by standard methods; therefore it seems likely that many of the relevant bacteria are not discovered in routine diagnostics, but may be relevant to pathogenesis. Culture-independent approaches such as NGS (Next generation Sequencing) have in principle made it possible to study or prove complex microbial colonization. Because NGS is a relatively new technology, microbiological diagnostic protocols need to be further customized and refined to integrate with the standard diagnostic workflow, if necessary. For microbiological diagnostics, material is collected from the appropriate ascites patients and sent for microbiological diagnostics. Afterwards the cultural diagnostics are carried out as part of the patient care at the university hospital. In this study the investigators plan to use these samples to analyze and compare the presence of bacteria by NGS in parallel to the culture diagnostics, and then compare it to the patients' gut microbiome, to understand the possible effect of the microbiome on ascites pathogenesis and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age
* Samples from patients who have ascites puncture to exclude infection
* Written consent of the patient after clarification

Exclusion Criteria:

* Minor patients
* Non-consenting patients
* Samples without sufficient residual material after standard diagnostics
* Samples from patients who have not consented to the examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult consent intensive care patients who undergo parenthesis for diagnostic purposes to exclude ascitic infection, regardless of the clinical picture. The indication for puncture is provided by the attending clinician regardless of the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The comparative assessment of about 50 patients | 12-18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tarek Badr, MD, Principal Investigator — Institute for Microbiology and Hygiene, Hermann-Herder-Str. 11, 79104 Freiburg
Locations (1):
- Institute for Microbiology and Hygiene, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided